CLINICAL TRIAL: NCT01045343
Title: Integrated Diagnostics Can Alter Heart Failure
Brief Title: Feasibility Study of an Integrated Diagnostic System to Manage Heart Failure
Acronym: INDICATE HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: INDICATE HF
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Heart Failure
Keywords: heart failure; home monitoring; integrated diagnostics; Cardiac Resynchronization Therapy with Defibrillator (CRT D)
MeSH Terms: conditions — Heart Failure | interventions — Office Visits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Active Comparator)
  Interventions: Other: Routine in office visits
- Integrated Diagnostics Arm (Experimental)
  Interventions: Other: Integrated diagnositic system

INTERVENTIONS:
Other: Integrated diagnositic system — Heart failure will be managed using the integrated diagnostic system which consists of patient tools and a new Heart Failure Clinician's website which displays a new Heart Failure Risk score. This Heart Failure Clinician's website will be reviewed every 2 weeks in addition to scheduled in-office visits every three months.
  Arms: Integrated Diagnostics Arm
Other: Routine in office visits — Heart failure will be managed with scheduled in-office visits every three months.
  Arms: Control Arm

SUMMARY:
The purpose of this clinical trial is to evaluate the potential benefits of a new heart failure diagnostic system for heart failure patients with implanted cardiac resynchronization therapy devices. This system consists of patient tools, a new heart failure risk score and a new clinician website. This study will evaluate this new system as a whole and establish the feasibility of implementing it into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide written informed consent
* Subject is at least 18 years of age
* Subject is willing and able to comply with the Clinical Investigation Plan
* Subject is currently enrolled in the Medtronic CareLink® Network
* Subject is currently a New Heart Association (NYHA) functional class III or NYHA functional class II with a heart failure related hospitalization within the past 180 days
* Subject has a Medtronic Concerto®/Consulta® cardiac resynchronization therapy (CRT)device implanted for at least 180 days
* Subject has been prescribed daily oral diuretic therapy for the management of heart failure

Exclusion Criteria:

* Subject is enrolled in a concurrent study with the exception of a study approved by the INDICATE HF Clinical Trial Leader
* Subject has a life expectancy of less than 1 year
* Subject's CRT device has an estimated battery life of less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change in subject self-care utilizing the Self-Care of Heart Failure Index | Baseline, 3 months, 6 months, 9 months
Proportion of time clinician and subject complied to protocol requirements for the new heart failure diagnostic system (patient tools and HF clinician website) | Baseline to 9 months
Number of clinical actions and types of health care utilizations in which actions are initiated | Baseline to 9 months
Subject outcomes including emergency room (ER) visits, hospitalization and death | Baseline to 9 months
Functional class using measurements including 6-minute hall walk and New York Heart Association class | Hall walk (Baseline to 9 months), NYHA (Baseline, 3 months, 6 months, 9 months)
Quality of life and depression scores utilizing measures including the Minnesota Living with Heart Failure Questionnaire and Patient Health Questionnaire | Baseline, 3 months, 6 months, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: INDICATE HF Team, Study Chair — Medtronic
Locations (13):
- United States (13):
  - Anchorage, Alaska
  - Aurora, Colorado
  - Tampa, Florida
  - Louisville, Kentucky
  - Jackson, Mississippi
  - Omaha, Nebraska
  - Voorhees Township, New Jersey
  - Cincinnati, Ohio
  - Abington, Pennsylvania
  - Doylestown, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Burlington, Vermont